CLINICAL TRIAL: NCT07393711
Title: Evaluation of the Effectiveness of Intrarenal Dioxidine Metaphylaxis for Preventing Recurrence of Infection Stones After Percutaneous Nephrolithotripsy
Brief Title: Metaphylaxis of Infected Kidney Stones After Percutaneous Nephrolithotripsy
Acronym: DIOX-PCNL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Kazakhstan Marat Ospanov Medical University (Other)
Responsible Party: Principal Investigator, Talgat A. Imzharov, Principal Investigator, West Kazakhstan Marat Ospanov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Approval No. 11 (11.16/03); EC Approval 11-16/03 (Other: Marat Ospanov Medical University)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Kidney Calculi; Nephrolithiasis; Urinary Tract Infections
Keywords: Percutaneous nephrolithotomy; PCNL; Infection stones; Struvite stones; Dioxidine; Intrarenal instillation; Stone recurrence; Metaphylaxis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urinary Tract Infections | interventions — dioxidine; Lithotripsy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive standard PCNL with or without adjunctive intrarenal dioxidine instillation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrarenal Dioxidine Group (Experimental): Participants undergo PCNL followed by intrarenal instillation of dioxidine to prevent infection-related stone recurrence.
  Interventions: Drug: Dioxidine; Procedure: Percutaneous Nephrolithotripsy (PCNL)
- Standard Treatment Group (Active Comparator): Participants undergo standard PCNL without adjunctive dioxidine.
  Interventions: Procedure: Percutaneous Nephrolithotripsy (PCNL)

INTERVENTIONS:
Drug: Dioxidine — Intrarenal instillation of dioxidine solution after PCNL to reduce bacterial colonization and prevent recurrence of infection-related stones.
  Other Names: Intrarenal Dioxidine Instillation; Dioxidine Solution
  Arms: Intrarenal Dioxidine Group
Procedure: Percutaneous Nephrolithotripsy (PCNL) — Standard percutaneous nephrolithotripsy procedure for removal of kidney stones.
  Other Names: PCNL; Percutaneous Stone Removal; Percutaneous Lithotripsy

SUMMARY:
Kidney stone recurrence, particularly infection-related stones, remains a significant clinical problem after percutaneous nephrolithotripsy (PCNL). Bacterial colonization and persistent infection are recognized contributors to stone recurrence.

This study evaluates the effectiveness of intrarenal dioxidine instillation as a metaphylactic measure to reduce recurrence of infection-related kidney stones following PCNL. Patients undergoing PCNL will receive standard treatment, with or without adjunctive intrarenal dioxidine administration. The study aims to assess whether this approach reduces stone recurrence and infection-related complications.

DETAILED DESCRIPTION:
Infection-related kidney stones are associated with urease-producing bacteria and carry a high risk of recurrence even after successful surgical removal. Percutaneous nephrolithotripsy (PCNL) is the standard treatment for large or complex renal calculi; however, residual infection and bacterial biofilms may contribute to recurrent stone formation.

Metaphylaxis strategies targeting infection control may reduce recurrence rates. Dioxidine is an antimicrobial agent with broad-spectrum activity against gram-positive and gram-negative bacteria and has been used locally in urological practice. Intrarenal instillation may help reduce bacterial colonization in the collecting system.

The purpose of this study is to evaluate the clinical effectiveness and safety of intrarenal dioxidine instillation as a metaphylactic intervention after PCNL for infection-related kidney stones. Outcomes include stone recurrence, urinary tract infection rates, and postoperative complications. The results may help define improved metaphylaxis strategies for patients with infection-related nephrolithiasis.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years

Patients undergoing percutaneous nephrolithotripsy (PCNL)

Infection-related kidney stones

Ability to provide written informed consent

Exclusion Criteria:

Age <18 years

Pregnancy or breastfeeding

Known hypersensitivity to dioxidine

Severe renal insufficiency or end-stage renal disease

Severe comorbid conditions that preclude participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of infection-related kidney stones | 12 months post-PCNL
  Proportion of patients with recurrent infection-related kidney stones within 12 months after percutaneous nephrolithotripsy, assessed by imaging studies (ultrasound or CT) and clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Bazylbek S Zhakiev, MD, Study Director — West Kazakhstan Marat Ospanov Medical University
Locations (1):
- West Kazakhstan Marat Ospanov Medical University, Aqtöbe, Kazakhstan

IPD SHARING:
Plan to Share IPD: No